CLINICAL TRIAL: NCT04608409
Title: A Phase I Dose-Escalation Study on the Safety of Lapatinib With Dose-Dense Paclitaxel in Patients With Platinum-Resistant Ovarian Cancer
Brief Title: Dose Escalation of Lapatinib With Paclitaxel in Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frederick R. Ueland, M.D. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Frederick R. Ueland, M.D., Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-GYN-06; 5P30CA177558-10 (NIH)
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
Keywords: platinum-resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Lapatinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lapatinib - Group 1 (Experimental): Patients in this group will receive Lapatinib (750mg PO BID) and Paclitaxel (80mg/m2).
  Interventions: Drug: Lapatinib and Paclitaxel
- Lapatinib - Group 2 (Experimental): Patients in this group will receive Lapatinib (1500mg PO BID) and Paclitaxel (80mg/m2).
  Interventions: Drug: Lapatinib and Paclitaxel
- Lapatinib - Group 3 (Experimental): Patients in this group will receive Lapatinib (2000mg PO BID) and Paclitaxel (80mg/m2).
  Interventions: Drug: Lapatinib and Paclitaxel

INTERVENTIONS:
Drug: Lapatinib and Paclitaxel — Participants will receive twice-daily Lapatinib, beginning two days prior to Paclitaxel treatment.

SUMMARY:
This trial will be a phase I dose-escalation study of lapatinib and paclitaxel for platinum-resistant ovarian cancer, which will establish the phase II dose for subsequent efficacy trials.

DETAILED DESCRIPTION:
While ABCB1 (P-glycoprotein 1) upregulation after paclitaxel administration is well known, there is currently no clinically available method for preventing or overcoming it. To develop a therapy able to prevent ABCB1 upregulation and paclitaxel resistance, several ABCB1 inhibitors have been evaluated in combination with paclitaxel in preclinical model systems. Pulsed-dose lapatinib and paclitaxel are synergistic and inhibition of ABCB1 by lapatinib increases sensitivity to paclitaxel. Lapatinib is FDA approved, orally available, and previously studied in combination with weekly paclitaxel for breast cancer at doses of 1000mg to 1250mg daily (7000-8250mg per week). This trial will use twice-daily dosing of lapatinib at a starting dose of 750 mg for 2 days (1500mg a day and 3000mg weekly dose), which is less than half of the continuous dose and has been shown to achieve plasma concentrations at 48 hours that are associated with synergy. Therefore, these findings can be translated into a novel, well-tolerated, and convenient combination regimen with significant potential for clinical activity. This trial will be a phase I dose-escalation study of lapatinib and paclitaxel for platinum-resistant ovarian cancer, which will establish the phase II dose for subsequent efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed ovarian cancer who recur within 12 months of platinum-based chemotherapy
* ECOG performance status less than or equal to 2
* Adequate organ and marrow function at baseline
* ability to sign a written informed consent document

Exclusion Criteria:

* hypersensitivity to lapatinib or paclitaxel
* uncontrolled intercurrent illness
* receiving medications that inhibit or induce CYP3A4
* malabsorption syndrome
* congestive heart failure
* receiving any other anti-cancer investigational agents
* baseline neuropathy greater than Grade 1

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Ueland, MD, Principal Investigator — Markey Cancer Center
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixteen patients were evaluable for efficacy, toxicity, and response.
Period: Overall Study
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3
Started | 3 | 6 | 7
Completed | 2 | 5 | 5
Not Completed | 1 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3 | Total
Number analyzed (Participants) | 3 | 6 | 7 | 16
Age, Continuous [Median (Full Range); unit: years] | 75 [72 to 79] | 64 [51 to 75] | 66 [53 to 70] | 67.5 [51 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 7 | 16
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 6 | 7 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival.
Description: Number of patients with progression-free survival at one year.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3
Number analyzed (Participants) | 3 | 6 | 7
Participants | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity
Description: Dose limiting toxicity (DLT) is calculated as the total number of patients experiencing DLTs divided by the total number treated.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3
Number analyzed (Participants) | 3 | 6 | 7
Participants | 0 | 1 | 1

3. Secondary Outcome: Change in Plasma Concentration of Lapatinib Cycle 1
Description: Plasma concentrations of lapatinib will be measured on days 8 and 15 prior to paclitaxel administration
Time Frame: 15 days (on day 8 and 15)
Population: Plasma lapatinib concentrations were analyzed among samples from patients who completed dosing for the assigned treatment arm and had blood drawn within 24 hours of the last lapatinib dose.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3
Number analyzed (Participants) | 3 | 4 | 4
ng/ml
  Day 8: number analyzed (Participants) | 3 | 4 | 3
  Day 8 | 2579 (1620) | 1593 (2100) | 2490 (1720)
  Day 15: number analyzed (Participants) | 2 | 4 | 4
  Day 15 | 1630 (590) | 2370 (1910) | 2851 (2160)

4. Other Pre Specified Outcome: ABCB1 Expression
Description: Levels of ABCB1 expression (cell-free RNA) will be measured using Nanostring sequencing.
Time Frame: 15 days (on day 1, 8 and 15)
Reporting Status: Not Posted

5. Secondary Outcome: Change in Plasma Concentration of Lapatinib Cycle 2
Description: Plasma concentrations of lapatinib will be measured on days 8 and 15 prior to paclitaxel administration
Time Frame: 15 days (on day 8 and 15)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3
Number analyzed (Participants) | 2 | 3 | 4
ng/ml
  Day 8 | 2002 (750) | 2987 (2900) | 2951 (2650)
  Day 15 | 2002 (1120) | 3393 (3940) | 2312 (1490)

6. Secondary Outcome: Change in Plasma Concentration of Lapatinib Cycle 3
Description: Plasma concentrations of lapatinib will be measured on days 8 and 15 prior to paclitaxel administration
Time Frame: 15 days (on day 8 and 15)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3
Number analyzed (Participants) | 2 | 3 | 4
ng/ml
  Day 8: number analyzed (Participants) | 1 | 2 | 4
  Day 8 | 1439 | 1499 (790) | 2175 (1790)
  Day 15 | 2242 (1460) | 1031 (600) | 1824 (1130)

ADVERSE EVENTS:
Time Frame: 30 days after discontinuation (last dose) of lapatinib, up to 3 cycles (a cycle is 28 days)
Description: If a participant experienced more than one adverse event within a toxicity category, the participant is counted once under that category. If a participant had more than one count for a particular toxicity, the participant was counted once for that toxicity.
  CTCAE v5.0 was used for coding.
Arm/Group | Lapatinib - Group 1 | Lapatinib - Group 2 | Lapatinib - Group 3
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/6 | 2/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib - Group 1 (N=3) | Lapatinib - Group 2 (N=6) | Lapatinib - Group 3 (N=7)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 | 0
Fever (General disorders) | 1 (1) | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 | 0
Platelet count decreased (Investigations) | 1 (1) | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib - Group 1 (N=3) | Lapatinib - Group 2 (N=6) | Lapatinib - Group 3 (N=7)
Lymphocyte count decreased (Investigations) | 2 (4) | 2 (3) | 5 (7)
White blood cell decreased (Investigations) | 2 (3) | 2 (4) | 5 (7)
Creatinine increased (Investigations) | 1 (4) | 3 (6) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 | 2 (3) | 1 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 | 2 (2)
Platelet count decreased (Investigations) | 1 (5) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 | 1 (1)
Other (Investigations) | 0 | 0 | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5) | 4 (8) | 4 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 5 (13)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 2 (3) | 5 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (8) | 3 (3) | 2 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 3 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 0 | 2 (4)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 5 (16) | 6 (22)
Nausea (Gastrointestinal disorders) | 0 | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 (2) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 | 5 (9) | 3 (9)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0
Fatigue (General disorders) | 0 | 2 (2) | 1 (1)
Fever (General disorders) | 1 (3) | 1 (1) | 0
Edema limbs (General disorders) | 0 | 1 (1) | 0
Gait disturbance (General disorders) | 0 | 0 | 1 (1)
Malaise (General disorders) | 0 | 1 (1) | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (3) | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 (2) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 2 (2) | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0
Other (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 1 (1) | 0
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0
Papulopustular rash (Infections and infestations) | 0 | 1 (1) | 0
Urinary tract infection (Infections and infestations) | 0 | 1 (1) | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 (2) | 0
Headache (Nervous system disorders) | 0 | 0 | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 (1) | 0
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0
Dysuria (Renal and urinary disorders) | 0 | 1 (1) | 0
Other (Renal and urinary disorders) | 0 | 1 (1) | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 (1) | 0
Other (Reproductive system and breast disorders) | 0 | 1 (1) | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1 (1) | 0
Flushing (Vascular disorders) | 0 | 1 (1) | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 (1) | 0
Insomnia (Psychiatric disorders) | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT04608409/Prot_SAP_ICF_000.pdf